CLINICAL TRIAL: NCT06873269
Title: Holmium-166 Transarterial Radioembolization for the Treatment of Hepatocellular Carcinoma
Acronym: TARE for HCC
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: TARE for HCC
Record Dates: First submitted 2025-02-21; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Hepatocellular Carcinoma; Liver Cirrhosis; Non-metastatic Hepatocellular Carcinoma
Keywords: holmium-166; transarterial radioembolization
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Baseline assessment — demographic information (age, gender, ethnicity), relevant medical, surgical and oncological history (number and types of previous treatments), clinical assessment (including Child Pugh score, BCLC stage), functional assessment (ECOG performance status), baseline laboratory findings (liver and kidney function, AFP tumor marker,..), date of diagnosis, baseline imaging characteristics (number, size, location of lesions, portal vein thrombosis, TNM stage) and if available histopathological diagnosis (grade of differentiation, microvascular invasion).
Radiation: holmium-166 radioembolization — Characteristics of treatment: treatment date, predicted target dose in Gy, predicted non-target dose in Gy, target volume in mL, whole liver volume in mL, administered activity in GBq, tumor absorbed dose, normal liver-absorbed dose Aim of TARE: palliative or curative/downstaging
Other: Follow-up phase — The following data on the performed monitoring after the procedure with clinical assessment, imaging modalities and blood samples as determined by the center, will be collected retrospectively:
  * Response: tumor response on imaging, tumor marker (AFP levels) at 3, 6 and 12 months after Ho166-TARE, and thereafter every 6 months until last follow-up or death, date of progression, time to progression after treatment
  * Toxicity and safety: side effects, adverse events, hepatic function parameters, presence of ascites or hepatic encephalopathy
  * Survival: date of last follow-up or death

SUMMARY:
This study aims to evaluate the effectiveness and safety of Holmium-166 (Ho-166) transarterial radioembolization (TARE) for treating patients with locally advanced hepatocellular carcinoma (HCC), a common type of liver cancer. HCC is often linked to conditions like liver cirrhosis and viral hepatitis, with a poor prognosis for advanced stages. TARE involves delivering radioactive particles directly to liver tumors, sparing healthy tissue and providing targeted radiation.

This study will include patients diagnosed with HCC who have received Holmium-166 TARE treatment between January 2010 and December 2024. Researchers will look at patient and tumor characteristics, side effects, how well the treatment works, and survival outcomes. The goal is to determine whether Holmium-166 TARE is a safe and effective treatment option for people with locally advanced HCC.

The findings will help doctors better understand how this therapy can be used to treat liver cancer and whether it can improve survival rates for patients with this challenging disease.

DETAILED DESCRIPTION:
This study investigates the use of Holmium-166 (Ho-166) transarterial radioembolization (TARE) as a treatment for patients with locally advanced hepatocellular carcinoma (HCC), a primary liver cancer. The research focuses on evaluating both the safety and effectiveness of this therapeutic approach in patients who have been diagnosed with HCC and treated with Ho-166 TARE between January 2010 and December 2024.

HCC is a highly aggressive cancer that commonly arises in individuals with liver cirrhosis, often due to underlying chronic viral hepatitis or metabolic dysfunction-associated fatty liver disease (MAFLD). As the disease progresses, treatment options become limited, particularly in cases where the cancer has reached advanced stages with symptoms, vascular invasion, or extrahepatic spread. Holmium-166 TARE is an interventional procedure that involves delivering microspheres containing the radioactive isotope Holmium-166 directly to the tumor site via the hepatic artery. This targeted radiation therapy is designed to maximize tumor destruction while minimizing damage to surrounding healthy liver tissue.

The study will retrospectively analyze the medical records of patients who received Ho-166 TARE as part of their treatment plan. This includes examining factors such as patient demographics, tumor characteristics, treatment-related side effects or toxicity, radiologic response to the therapy, progression-free survival (PFS), and overall survival (OS). The primary aim is to assess whether Ho-166 TARE provides a significant benefit in terms of tumor response, survival outcomes, and safety when compared to other treatment modalities.

Pre-treatment planning for Holmium-166 TARE involves a detailed assessment of the liver's blood supply through angiography and the use of cone-beam CT and SPECT/CT scans to guide precise delivery of the radioactive microspheres. The dosage is tailored to each patient, aiming to deliver over 150 Gy to the tumor while keeping the healthy liver dose below critical thresholds.

By focusing on a diverse patient population with locally advanced HCC, this study seeks to provide important data that could help refine treatment strategies for liver cancer. The results may support the broader use of Ho-166 TARE in clinical practice, especially for patients who are not eligible for curative treatments like surgery or liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 year or older
* diagnosed with locally advanced HCC without extra-hepatic metastases
* HCC must not be amendable to treatment by surgical resection or percutaneous radiofrequency ablation
* after assessment by the investigator and multidisciplinary tumor board, the patient is considered suitable for protocol treatment with Holmium-166 TARE
* ECOG performance status 0-2
* child-Pugh A-B
* tumor response evaluable with mRECIST criteria during follow-up

Exclusion Criteria:

* prior treatment with any of the following treatment modalities for HCC: systemic therapy, hepatic radiation therapy
* currently enrolled in clinical studies where patient receive investigational therapeutic drug
* metastatic disease
* concurrent malignancy
* active contra-indications to angiography or selective catherization (i.e. severe vascular disease or bleeding diathesis)
* uncontrolled and/or severe comorbidities (active infection, heart failure,...) with limited estimated life expectancy
* history of or know allergic reactions to used compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients must have been diagnosed with HCC based on:
     o Mass larger than 1 cm with pathognomonic HCC imaging hallmarks (arterial phase hyperenhancement (APHE) and washout on portal venous and/or delayed phases) on multiphasic contrast-enhanced CT or MRI in a cirrhotic liver.
     AND/OR
     o Lesions in the liver with histopathological diagnosis of HCC on biopsy.
  2. Based on BCLC staging, the disease must be locally advanced without extra-hepatic disease and after assessment by a multidisciplinary tumor board, the patient was considered suitable for protocol treatment with Holmium-166 TARE
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
efficacy of Holmium-166 TARE in patients with locally advanced HCC | through study completion, on average 60 months
  To assess the efficacy of Holmium-166 TARE in patients with locally advanced HCC in terms of tumor response rate (RR)
efficacy of Holmium-166 TARE in patients with locally advanced HCC | through study completion, on average 60 months
  To assess the efficacy of Holmium-166 TARE in patients with locally advanced HCC in terms of overall survival (OS)

SECONDARY OUTCOMES:
progression-free survival (PFS), time to disease progression and toxicity and safety during follow-up | through study completion, on average 60 months
  progression-free survival (PFS), time to disease progression and toxicity and safety during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided